CLINICAL TRIAL: NCT06637527
Title: A Phase 2a, Randomized, Double-Masked, Placebo-Controlled Study Assessing the Safety and Efficacy of OK-101 Treatment in Subjects With Neuropathic Corneal Pain
Brief Title: The Study Assessing the Safety and Efficacy of OK-101 Treatment in Subjects With Neuropathic Corneal Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study ended early to expedite development and enable earlier FDA discussions. Prior Phase 2 data (240 patients) showed favorable safety and placebo-like tolerability. Closure was not due to safety concerns.
Sponsor: Okyo Pharma Ltd (Industry)
Collaborators: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: OK-101-NCP-001-23
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-10

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Approximately 48 subjects will be randomized in a 1:1:1 ratio to receive treatment with 0.05% OK-101 (Arm A) or 0.1% OK-101 (Arm B) or placebo (Arm C).
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a randomized, double-masked, placebo-controlled trial to investigate the efficacy of OK101 study drug in treating the symptoms of NCP at baseline (Visit 1) through the end of study (16 weeks) in NCP subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (Experimental): OK-101, 0.05% - one drop of study drug (0.05%) will be instilled in affected eye(s), four times daily (every 4 hours up to 16 hours, e.g., 9:00 am, 01:00 pm; 05:00 pm, 09:00pm) for 12 weeks
  Interventions: Drug: OK-101 0.05%
- Arm B (Experimental): OK-101, 0.1% - one drop of study drug (0.1%) will be instilled in affected eye(s), four times daily (every 4 hours up to 16 hours, e.g., 9:00 am, 01:00 pm; 05:00 pm, 09:00pm) for 12 weeks.
  Interventions: Drug: OK-101 0.1%
- Arm C (Placebo Comparator): Placebo - one drop of placebo will be instilled in affected eye(s), four times daily (every 4 hours up to 16 hours, e.g., 9:00 am, 01:00 pm; 05:00 pm, 09:00pm) for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OK-101 0.05% — 0.05% Ophthalmic Solution
  Arms: Arm A
Drug: OK-101 0.1% — 0.1% Ophthalmic Solution
  Arms: Arm B
Drug: Placebo — Placebo
  Arms: Arm C

SUMMARY:
The primary objective of this study, in subjects with Neuropathic Corneal Pain, is to evaluate the efficacy and safety of OK-101 0.05% and 0.1% as compared to placebo instilled 4 times/day in subjects with neuropathic corneal pain, as assessed by visual analogue scale (VAS).

DETAILED DESCRIPTION:
Detailed Description: Neuropathic corneal pain (NCP) is a complex disease affecting the somatosensory nervous system characterized by different underlying etiologies and pathogenesis.

OK-101 is a lipid conjugated chemerin peptide antagonist of the ChemR23 G-protein coupled receptor which is typically found on immune cells of the eye responsible for the inflammatory response. OK-101 has been shown to produce anti-inflammatory and pain-reducing activities in mouse models of dry eye disease and neuropathic corneal pain; and is designed to combat washout through the inclusion of the lipid 'anchor' contained in the candidate drug molecule to enhance the residence time of OK-101 within the ocular environment. Our preclinical studies have shown that treatment with OK-101 abolishes corneal pain in a murine model of NCP.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years.
2. Symptoms of neuropathic corneal pain for at least 3 months, such as burning, stinging, light sensitivity, discomfort, or pain.
3. Positive IVCM findings evaluated by an experienced ophthalmologist (Pedram Hamrah, M.D.): decreased nerve density AND evidence of microneuromas.
4. Females of childbearing potential must have a negative pregnancy test.
5. Best corrected distance visual acuity (BCDVA), using corrective lenses, if necessary, in the study eye of at least +1.0 Log MAR (Snellen <20/200).
6. Satisfying all Informed Consent requirements.
7. Ability and willingness to comply with study procedures.

Exclusion Criteria:

1. Evidence of any active ocular infection.
2. Evidence of any intraocular inflammation.
3. Evidence of any persistent epithelial defect/ulcer.
4. Evidence of any corneal scar/corneal edema.
5. Presence of any other ocular conditions that require topical medications during the treatment phase.
6. History of severe systemic allergy or severe ocular allergy.
7. Inability to suspend topical medications 8 days prior to the starting date.
8. Inability to continue oral medications for NCP without changes during the study duration.
9. No changes or less than 50% improvement in VAS score after topical 0.5% proparacaine hydrochloride (Alcaine, Alcon, Fort Worth, TX).
10. History of any ocular surgery within three months before study Visit 1(day 0).
11. Ocular surgery expected during the 16 weeks of the trial.
12. Use of refractive/therapeutic contact lenses during the study period.
13. Female subjects who are pregnant/have a positive pregnancy test result or are breastfeeding or intend to become pregnant during the study treatment period.
14. Drug addiction/alcohol abuse within the last year.
15. Participation in another clinical trial concurrently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Assess ocular pain using 0-10 visual analog scale (VAS) | 16 Weeks
  Visual analog scale questionaire will be used to evaluate the pain on 0-10 scale where 0 is no pain and 10 is worst pain imaginable.

SECONDARY OUTCOMES:
Ocular Pain Assessment Survey (OPAS) scores | 16 Weeks
  Twenty-seven item questionnaires specifically designed to assess symptoms and quality of life in ocular pain.
Ocular Surface Disease Index (OSDI©) scores | 16 Weeks
  Twelve-item questionnaire to assess symptoms of ocular irritation consistent with dry eye and their impact on vision-related functioning.
QoL Improvement assesed by OPAS score | 16 Weeks
  Twenty-seven item questionnaires specifically designed to assess symptoms and quality of life in ocular pain
Drop comfort Scores | 16 Weeks
  Drop Comfort will be assesed using Scale 0-10, with a value of 0 being most comfortable and 10 being least comfortable.

OTHER OUTCOMES:
Asses corneal sensitivity thresholds obtained with the Cochet Bonnet esthesiometer on 0-6 scale (in cm) | 16 Weeks
  Corneal Sensitivity will be measured using a Cochet Bonnet aesthesiometer before the instillation of any dilating or anesthetic eye drops. Corneal sensitivity will be assessed in the qualifying NEI zones of each eye. This instrument is constituted by a retractable 6 cm length filament of 0.12 mm in diameter, and it is considered the gold standard for corneal sensation assessment. We will gently press the monofilament against the cornea, and we will shorten it in steps of 1.0 cm if a negative response is obtained. If a positive response is obtained, we will advance the monofilament by 0.5cm, and we will consider the corneal sensitivity as the longest filament length necessary to obtain a positive response.
Asses corneal nerve regeneration by measuring change in total length of corneal nerve regeneration | 16 Weeks
  Change in total length of all nerves within an image (in mm/mm2) will be evaulated via In-Vivo Confocal Microscopy (IVCM) imaging
Assess change in numbers of microneuromas | 16 Weeks
  Presence of microneuromas will be graded from In-Vivo Confocal Microscopy (IVCM) imaging
Asses change in dendritiform cells density by In-Vivo Confocal Microscopy (IVCM) imaging | 16 Weeks
  Change in dendritiform cells density (in cells/mm^2) of Corneal Immune Dendritiform Cells will be assesed via Via In-Vivo Confocal Microscopy (IVCM) imaging

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States